CLINICAL TRIAL: NCT01663766
Title: A Phase I Study of Milatuzumab (hLL1) for Prevention of Acute Graft Versus Host Disease Following Reduced-Intensity Conditioning Allogeneic Stem Cell Transplant in Patients With Hematologic Malignancies
Brief Title: Phase I Study of Milatuzumab for Graft Versus Host Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PIs agreed no safety signals were shown, drug did not appear to lessen the risk of preventing GVHD no further patients would be enrolled
Sponsor: Gilead Sciences (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-IMMU-115-03
Record Dates: First submitted 2012-08-07; First posted 2012-08-13 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2020-09

CONDITIONS: GVHD (Acute or Chronic); Acute Myeloid or Lymphoblastic Leukemia (AML or ALL); Myelodysplastic Syndrome; Chronic Myelogenous Leukemia (CML); Multiple Myeloma (MM); Non-Hodgekin Lymphoma (NHL-both Follicular & Diffuse Large Cell); Chronic Lymphocytic Leukemia or Small Lymphocytic Leukemia (CLL or SLL)
Keywords: GVHD (acute or chronic); acute myeloid or lymphoblastic leukemia (AML or ALL); myelodysplastic syndrome; Chronic myelogenous leukemia (CML); Multiple Myeloma (MM); Non-Hodgekin lymphoma (NHL-both follicular & diffuse large cell); Chronic lymphocytic leukemia or small lymphocytic leukemia (CLL or SLL)
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milatuzumab (Experimental): Milatuzumab will be added to the standard GVHD reduced intensity consitioning and prophylaxis regimen of fludarabine, busulfan, tacrolimus and low-dose methotrexate.
  Interventions: Drug: milatuzumab

INTERVENTIONS:
Drug: milatuzumab — Milatuzumab is a humanized anti-CD74 antibody that is administered intravenously.
  Other Names: IMMU-115; hLL1; anti-CD74

SUMMARY:
This study will assess the safety and tolerability of milatuzumab (IMMU-115) when added to a standard regimen to prevent Graft vs. Host Disease (GVHD) in patients with hematologic malignancies undergoing stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females, ≥ 18 years of age
* Able to understand and willing to sign informed consent.
* Histologically confirmed hematologic malignancy that is deemed best treated by RIC allogeneic SCT, including:
* Acute myeloid or lymphoblastic leukemia (AML, ALL) with < 5% blasts in the bone marrow
* Myelodysplastic syndrome and intermediate-2 or high-risk IPSS score with < 5% blasts in the bone marrow
* Chronic myelogenous leukemia failing to respond to at least two different tyrosine kinase inhibitors
* Multiple myeloma that has relapsed following autologous stem cell transplant
* Follicular lymphoma (grades 1, 2, or 3a by WHO criteria) or monocytoid lymphoma that has relapsed following at least two prior chemotherapy regimens and with either no lymph node groups ≥ 3 cm or with a ≥ 50% reduction in estimated lymph node diameter with most recent salvage therapy
* Diffuse large B-cell NHL that has relapsed after at least 2 prior chemotherapy regimens (could include high-dose chemotherapy with autologous stem cell rescue) and is still sensitive to chemotherapy by virtue of a PR or CR following most recent salvage chemotherapy
* Transformed follicular lymphoma that has achieved a PR or CR following chemotherapy
* Mantle cell lymphoma that has relapsed after at least 2 prior chemotherapy regimens (could include high-dose chemotherapy with autologous stem cell rescue)
* CLL/SLL/PLL that meets one of the following:
* del (17p13.1) in first remission
* Response no better than a PR with chemoimmunotherapy or relapse within 2 years of chemoimmunotherapy
* Richter's transformation
* Complex karyotype
* At least 4 weeks beyond prior chemotherapy (excluding steroids), antibody therapy, radiation, or radioimmunoconjugate therapy, and with any kinase inhibitors discontinued at least one week prior to starting the conditioning regimen.
* ECOG performance status ≤ 2
* Life expectancy of greater than 3 months
* Adequate organ function measured by the following within seven days of beginning conditioning:
* AST (SGOT) ≤ 3.0 x institutional upper limit of normal (IULN)
* Total bilirubin ≤ 1.5 xIULN unless due to Gilbert's disease
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 50 mL/min
* DLCO > 40% with no symptomatic pulmonary disease
* LVEF by echocardiogram or MUGA of at least 30%
* Women of child bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
* Matched (8/8) related or matched unrelated donor identified. Haploidentical or umbilical cord grafts are not allowed.
* Donor willing to donate peripheral blood stem cells and meets institutional criteria for stem cell donation.

Exclusion Criteria:

* Prior allogeneic stem cell transplant
* Patients requiring a myeloablative conditioning regimen
* Patients best served by a bone marrow transplant are not eligible as this study will be restricted only to peripheral stem cells.
* No suitable donor identified
* Prior anaphylactic response or Grade 4 infusion reaction to milatuzumab
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active hepatitis B infection are not eligible. Patients with a history of hepatitis B (surface antigen or core antibody positive) must take lamivudine or equivalent during study therapy and for one year after completion of milatuzumab.
* LVEF < 30%
* Seropositivity for HIV or Hepatitis C
* Patients with known CNS lymphoma are excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Active secondary malignancies with the exception of non-melanomatous skin cancers or low risk prostate cancer under observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
All patients administered any dose of study drug will be included in the evaluation of safety | Safety will be assessed by measuring the change from baseline during 7 days of treatment and up to 30 days after treatment
  Safety will be measured by physical examinations and hematology and chemistry blood tests. Cardiac safety will be done using MUGA scans or echocardiograms. These assessments will be done routinely during treatment and up to 30 days after treatment and any change from baseline will be assessed. Long term safety will be assessed every 3 months after that for up to 1 year; any change from baseline will be assessed.

SECONDARY OUTCOMES:
Determine the therapeutic efficacy of milatuzumab in this patient population | Efficacy will be assessed 30 days after treatment.
  Acute GVHD will be assessed at days +30 and +100 by laboratory testing. Chronic GVHD assessment will be performed at days +100, +270 & +365 after stem cell transplant.

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States